CLINICAL TRIAL: NCT02202525
Title: Evolution of Pulse Pressure Following Initiation of Antihypertensive Therapy
Brief Title: Evolution of Pulse Pressure Following Initiation of Antihypertensive Therapy in Patients With Essential Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.362
Record Dates: First submitted 2014-07-28; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Essential arterial hypertension: Patients with essential arterial hypertension needing a new antihypertensive therapy
  Interventions: Drug: Micardis®; Drug: Other hypertensives

INTERVENTIONS:
Drug: Micardis®
  Other Names: Telmisartan
Drug: Other hypertensives

SUMMARY:
The main purpose of this prospective, multicentre, french observational study is to analyse the evolution of pulse pressure (PP) and to identify its prognostic factors in hypertensive patients three months after initiation of a new hypertensive therapy. The PP is defined as the difference between systolic blood pressure (SBP) and diastolic blood pressure (DBP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential arterial hypertension needing a new antihypertensive therapy
* A patient was included by the physician only if he/she had agreed after being informed about the study

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with essential hypertenstion treated by private or hospital cardiologists
Sampling Method: Non-Probability Sample
Enrollment: 2148 (Actual)
Dates: Start 2001-01; Primary Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in pulse pressure | Up to 3 months after start of treatment
Number of patients with adverse drug reactions | Up to 3 months after start of treatment